CLINICAL TRIAL: NCT05559138
Title: Analysis of Clinical Characteristics of Hemodialysis Patients With Omicron Infection
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IIT-2022-0120
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
Keywords: hemodialysis
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hemodialysis patients with omicron infection: hemodialysis patients with omicron infection
  Interventions: Other: no intervention
- non-hemodialysis patients with omicron infection: non-hemodialysis patients with omicron infection
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
By collecting the clinical data of hemodialysis patients with Omicron infection in RenJi Hospital from April 7, 2022 to June 10, 2022, the clinical characteristics of this population were analyzed. And to analyze the risk factors of different clinical outcomes according to the clinical outcome of this population.

DETAILED DESCRIPTION:
This study was a single-center, retrospective, observational study. The research subjects were hemodialysis patients admitted to the Hemodialysis Center of Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine because of omicron infection during the Omicron epidemic period from April 7, 2022 to June 10, 2022. 65 cases were included in the study after excluding those patients who underwent hemodialysis due to acute kidney injury. And they were compared with 195 non-dialysis patients admitted to the hospital in the same period,who were randomly selected, according to the ratio of 1:3.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patients due to chronic kidney disease stage 5 with omicron infection

Exclusion Criteria:

* Patients on hemodialysis due to acute kidney injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with omicron infection
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Viral elimination | 2022-4-7 to 2022-6-10
  both negative for ORF1ab and N genes (Ct value ≥35 by real-time PCR) in two consecutive days.

SECONDARY OUTCOMES:
cardiovascular events | 2022-4-7 to 2022-6-10
  including acute left heart failure, new symptomatic arrhythmias requiring drug control, acute coronary syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Jiayue Lu, Study Director — Renji Hospital affiliation to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Result] De Meester J, De Bacquer D, Naesens M, Meijers B, Couttenye MM, De Vriese AS; NBVN Kidney Registry Group. Incidence, Characteristics, and Outcome of COVID-19 in Adults on Kidney Replacement Therapy: A Regionwide Registry Study. J Am Soc Nephrol. 2021 Feb;32(2):385-396. doi: 10.1681/ASN.2020060875. Epub 2020 Nov 5. PMID 33154174
- [Result] Shuai H, Chan JF, Hu B, Chai Y, Yuen TT, Yin F, Huang X, Yoon C, Hu JC, Liu H, Shi J, Liu Y, Zhu T, Zhang J, Hou Y, Wang Y, Lu L, Cai JP, Zhang AJ, Zhou J, Yuan S, Brindley MA, Zhang BZ, Huang JD, To KK, Yuen KY, Chu H. Attenuated replication and pathogenicity of SARS-CoV-2 B.1.1.529 Omicron. Nature. 2022 Mar;603(7902):693-699. doi: 10.1038/s41586-022-04442-5. Epub 2022 Jan 21. PMID 35062016
- [Result] Halfmann PJ, Iida S, Iwatsuki-Horimoto K, Maemura T, Kiso M, Scheaffer SM, Darling TL, Joshi A, Loeber S, Singh G, Foster SL, Ying B, Case JB, Chong Z, Whitener B, Moliva J, Floyd K, Ujie M, Nakajima N, Ito M, Wright R, Uraki R, Warang P, Gagne M, Li R, Sakai-Tagawa Y, Liu Y, Larson D, Osorio JE, Hernandez-Ortiz JP, Henry AR, Ciuoderis K, Florek KR, Patel M, Odle A, Wong LR, Bateman AC, Wang Z, Edara VV, Chong Z, Franks J, Jeevan T, Fabrizio T, DeBeauchamp J, Kercher L, Seiler P, Gonzalez-Reiche AS, Sordillo EM, Chang LA, van Bakel H, Simon V; Consortium Mount Sinai Pathogen Surveillance (PSP) study group; Douek DC, Sullivan NJ, Thackray LB, Ueki H, Yamayoshi S, Imai M, Perlman S, Webby RJ, Seder RA, Suthar MS, Garcia-Sastre A, Schotsaert M, Suzuki T, Boon ACM, Diamond MS, Kawaoka Y. SARS-CoV-2 Omicron virus causes attenuated disease in mice and hamsters. Nature. 2022 Mar;603(7902):687-692. doi: 10.1038/s41586-022-04441-6. Epub 2022 Jan 21. PMID 35062015
- [Result] Lewnard JA, Hong VX, Patel MM, Kahn R, Lipsitch M, Tartof SY. Clinical outcomes associated with SARS-CoV-2 Omicron (B.1.1.529) variant and BA.1/BA.1.1 or BA.2 subvariant infection in Southern California. Nat Med. 2022 Sep;28(9):1933-1943. doi: 10.1038/s41591-022-01887-z. Epub 2022 Jun 8. PMID 35675841